CLINICAL TRIAL: NCT05629923
Title: EVALUATION OF COVID-19 VACCINATION EFFICACY AND CONTIXAGEVIMAB-CILGAVIMAB PROPHYLAXIS IN LIVER AND KIDNEY TRANSPLANT PATIENTS: PRELIMINARY STUDY
Brief Title: EVALUATION OF DIFFERENT PROPHYLACTIC INTERVENTIONS TOWARD COVID-19 IN SOLID ORGAN TRANSPLANT PATIENTS
Status: Completed | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Roberta Angelico, Lecturer in General Sugery PhD FEBS, University of Rome Tor Vergata
Other Study IDs: COVID-19 TRANPLANT
Record Dates: First submitted 2022-11-27; First posted 2022-11-29 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: COVID-19 Pandemic; Transplant-Related Disorder
Keywords: transplant; Vaccination; COVID-19 pandemic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Kidney and Liver Transplant: All Kidney and Liver Transplant recipients who are at follow-up in our institution will be enrolled. anti-COVID-19 title was obtained by ECLIA Test(Elyx, Roche). In the case of antibody level <100 IU/ml, patients were invited to prophylaxis with tixagevimab-cilgavimab(AZD7442, AstraZeneca). At three months, a follow-up was performed to assess any COVID-19 infection.
  Interventions: Drug: tixagevimab-cilgavimab(AZD7442, AstraZeneca)

INTERVENTIONS:
Drug: tixagevimab-cilgavimab(AZD7442, AstraZeneca) — In the case of antibody level <100 IU/ml, patients were invited to prophylaxis with tixagevimab-cilgavimab(AZD7442, AstraZeneca).

SUMMARY:
The goal of this observational study is to evaluate the immune response after COVID-19 vaccination in Liver(LT) and Kidney(KT) transplant recipient. The main question it aims to answer are:

* the evaluation of the antibody response after complete vaccination
* the efficacy of prophylaxis with long-acting-antibody prophylaxis (LAAB)

All LT and KT patients during follow-up have been enrolled. anti-COVID-19 title was obtained by Electrochemiluminescence Immunoassay (ECLIA) Test(Elyx, Roche). In the case of antibody level <100 IU/ml, patients were invited to prophylaxis with tixagevimab-cilgavimab(AZD7442, AstraZeneca). At three months, a follow-up was performed to assess any COVID-19 infection. At Six months another anti-COVID-19 title is obtained by ECLIA Test(Elyx, Roche) in LT and KT who undergo to LAAB.

DETAILED DESCRIPTION:
Liver(LT) and kidney(KT) transplant patients are at high risk of mortality from COVID-19(16-29%, 28%; respectively). Although transplant patients undergo a full vaccination course(3 doses), they are frequently low-responders and long-acting-antibody prophylaxis (LAAB) has been proposed. However, the efficacy of these strategies has not yet been demonstrated in LT and KT.

The goal of this observational study is to evaluate the immune response after COVID-19 vaccination in Liver(LT) and Kidney(KT) transplant recipient. The main question it aims to answer are:

* the evaluation of the antibody response after complete vaccination
* the efficacy of prophylaxis with long-acting-antibody prophylaxis (LAAB)

All LT and KT patients during follow-up have been enrolled. anti-COVID-19 title was obtained by Electrochemiluminescence Immunoassay (ECLIA) Test(Elyx, Roche). In the case of antibody level <100 IU/ml, patients were invited to prophylaxis with tixagevimab-cilgavimab(AZD7442, AstraZeneca). At three months, a follow-up was performed to assess any COVID-19 infection. At Six months another anti-COVID-19 title is obtained by ECLIA Test(Elyx, Roche) in LT and KT who undergo to LAAB.

ELIGIBILITY:
Inclusion Criteria:

* KT and LT transplant patients in follow up in Tor Vergata University
* Age >18 years
* At least 3 month post transplantation

Exclusion Criteria:

* pediatric recipients
* Active covid infection at the time of the study
* Pregnancy
* Allergy to any ingredients included in the vaccine
* Acute liver or kidney acute rejection proven by biopsy
* Acute Febrile state with either leucopenia or leucocytosis
* High dose of corticosteroid at study timing (pulse methyl prednisolone)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent KT and LT transplant currently in follow up in Tor Vergata University hospital
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
COVID-19 vaccination response rate | time 0
  The objective of our study is the evaluation of the antibody response after complete vaccination. The anti-COVID-19 title was obtained by ECLIA Test(Elyx, Roche).
Clinical efficacy of LAAB prophylaxis | three months from LAAB prophilaxys
  After COVID-19 title evaluation, in the case of antibody level <100 IU/ml, patients were invited to prophylaxis with tixagevimab-cilgavimab(AZD7442, AstraZeneca). At three months, a follow-up was performed to assess any COVID-19 infection.

SECONDARY OUTCOMES:
Serological title at six months | Six months from LAAB prophylaxis
  At six months, all the patients who underwent to to prophylaxis with tixagevimab-cilgavimab(AZD7442, AstraZeneca), the anti-COVID-19 title was obtained by ECLIA Test(Elyx, Roche).

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi di Roma Tor Vergata, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hardgrave H, Wells A, Nigh J, Klutts G, Krinock D, Osborn T, Bhusal S, Rude MK, Burdine L, Giorgakis E. COVID-19 Mortality in Vaccinated vs. Unvaccinated Liver & Kidney Transplant Recipients: A Single-Center United States Propensity Score Matching Study on Historical Data. Vaccines (Basel). 2022 Nov 13;10(11):1921. doi: 10.3390/vaccines10111921. PMID 36423017
- [Background] Angelico R, Blasi F, Manzia TM, Toti L, Tisone G, Cacciola R. The Management of Immunosuppression in Kidney Transplant Recipients with COVID-19 Disease: An Update and Systematic Review of the Literature. Medicina (Kaunas). 2021 Apr 30;57(5):435. doi: 10.3390/medicina57050435. PMID 33946462
- [Background] Levin MJ, Ustianowski A, De Wit S, Launay O, Avila M, Templeton A, Yuan Y, Seegobin S, Ellery A, Levinson DJ, Ambery P, Arends RH, Beavon R, Dey K, Garbes P, Kelly EJ, Koh GCKW, Near KA, Padilla KW, Psachoulia K, Sharbaugh A, Streicher K, Pangalos MN, Esser MT; PROVENT Study Group. Intramuscular AZD7442 (Tixagevimab-Cilgavimab) for Prevention of Covid-19. N Engl J Med. 2022 Jun 9;386(23):2188-2200. doi: 10.1056/NEJMoa2116620. Epub 2022 Apr 20. PMID 35443106